CLINICAL TRIAL: NCT00458796
Title: Cost-Effective Use of Bisphosphonates in Metastatic Bone Disease - A Comparison of Bone Marker Directed Zoledronic Acid Therapy to a Standard Schedule
Brief Title: Comparison of Two Schedules of Zoledronic Acid in Treating Patients With Breast Cancer That Has Spread to the Bone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lower than expected recruitment
Sponsor: University of Leeds (Other)
Collaborators: University of Sheffield (Other)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000538879; NCRI-BISMARK; ISRCTN83586728; EU-20716; EUDRACT-2005-001376-12
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Hypercalcemia of Malignancy; Metastatic Cancer; Musculoskeletal Complications; Pain
Keywords: hypercalcemia of malignancy; musculoskeletal complications; pain; stage IV breast cancer; male breast cancer; recurrent breast cancer; bone metastases
MeSH Terms: conditions — Breast Neoplasms; Humoral Hypercalcemia Of Malignancy; Neoplasm Metastasis; Pain; Breast Neoplasms, Male | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Zoledronic acid may help decrease the risk of broken bones, bone pain, and other symptoms caused by bone metastases. It may also help patients live more comfortably.

PURPOSE: This randomized clinical trial is studying different schedules of zoledronic acid to compare how well they work in treating patients with breast cancer that has spread to the bone.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the frequency and timing of serious related events (e.g., fractures, radiotherapy to bone, hypercalcemia of malignancy, orthopedic surgery, and spinal cord compression) in patients with advanced breast cancer metastatic to the bone treated with bone marker-directed schedule vs standard schedule zoledronic acid.

Secondary

* Compare the quality of life of patients treated with these regimens.
* Compare the clinical burden of skeletal complications in these patients.
* Compare pain, performance status, and analgesic use (PPA score) in these patients.
* Compare the incidence of new bone metastases in these patients.
* Compare overall survival of these patients.
* Compare bisphosphonate use and expenditure on administration in these patients.

OUTLINE: This is an open-label, randomized, controlled, parallel-group, multicenter study. Patients are stratified according to treatment center, gender, type of concurrent systemic therapy at study entry (endocrine therapy [with or without trastuzumab (Herceptin^®)] vs chemotherapy [with or without trastuzumab] vs trastuzumab alone vs chemotherapy and endocrine therapy [with or without trastuzumab] vs no systemic anticancer treatment), prior skeletal-related event (yes vs no), duration of bisphosphonate use for metastatic disease prior to study entry (4-6 months vs 6-12 months), type of metastases present at study entry (bone only vs bone and soft tissue vs bone and visceral metastases vs bone, soft tissue, and visceral metastases). Patients are randomized to 1 of 2 treatment arms.

* Arm I (standard schedule): Patients receive zoledronic acid IV over 15 minutes once every 3-4 weeks for 24 months.
* Arm II (bone marker-directed schedule): Patients receive zoledronic acid IV over 15 minutes once every 3-4, 8-9, or 15-16 weeks (based on serum N-telopeptide:creatinine ratio) for 24 months.

Quality of life is assessed at baseline and at 3, 6, 9, 12, 18, and 24 months.

After completion of study therapy, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 1,500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary breast cancer

  * Advanced disease
* Radiographic confirmation of bone metastases (≥ 1 bone scan lesion must be confirmed as metastatic by plain radiographs or CT scan/MRI)

  * Must have received zoledronic acid to treat metastatic bone disease (i.e., ≥ 4 or 5 zoledronic acid treatments prior to study entry for patients receiving 4- or 3-weekly infusions, respectively) for ≥ 4 months prior to study entry
  * Any bisphosphonate to treat metastatic bone disease allowed provided it was not given for more than 12 months prior to study entry
* No metabolic bone disease (e.g., Paget's disease of bone)

  * Osteoporosis allowed
* No brain metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* WHO or ECOG performance status 0-2
* Life expectancy ≥ 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine clearance ≥ 30 mL/min
* No poor venous access
* No concurrent active dental problems, including infection of the teeth or jawbone (maxilla or mandibular)
* No prior or current diagnosis of osteonecrosis of the jaw
* No other cancer within the past 5 years except nonmelanomatous skin cancer, carcinoma in situ of the uterine cervix, or superficial bladder cancer treated with curative intent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other prior bisphosphonate treatment within the past 3 weeks
* No treatment with systemic bone-seeking radioisotopes (e.g., strontium chloride Sr 89, samarium Sm 153 lexidronam pentasodium) within the past 3 months
* No wide-field (hemibody) radiotherapy within the past 3 months

  * Recent standard-field, localized radiotherapy allowed
* No dental or jaw surgery (e.g., extractions, implants) within the past 4 weeks
* No other concurrent bisphosphonates
* No concurrent medication with drugs known to affect bone metabolism (e.g., calcitonin or high-dose systemic corticosteroids [> 10 mg prednisolone/day or equivalent])

  * Systemic or oral corticosteroids allowed for clearly indicated conditions (e.g., chemotherapy-induced emesis, brain metastases, compression syndromes)
* Concurrent chemotherapy, biological therapy, or endocrine therapy allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2006-03

PRIMARY OUTCOMES:
Fractures
Radiotherapy to bone either for relief of pain or to treat or prevent pathological fractures or spinal cord compression
Hypercalcemia of malignancy
Orthopedic surgery to prevent or treat pathological fractures or spinal cord compression
Spinal cord compression

SECONDARY OUTCOMES:
Quality of life as measured by QLQ-C30 and the QLQ-BR23 breast-specific module
Clinical burden of skeletal complications
Pain, performance status, and analgesic use
Incidence of new bone metastases
Overall survival
Bisphosphonate use and expenditure on administration
Health care utilization
Clinical utility of the "point of care" test for N-telopeptides (NTx) excretion

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Coleman, MD, FRCP, Study Chair — Cancer Research Centre at Weston Park Hospital
Locations (30):
- United Kingdom (30):
  - Royal Bournemouth Hospital, Bournemouth, England
  - Derbyshire Royal Infirmary, Derby, England
  - Doncaster Royal Infirmary, Doncaster, England
  - University Hospital of North Durham, Durham, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Christie Hospital, Manchester, England
  - Withington Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - George Eliot Hospital, Nuneaton, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Solihull Hospital, Solihull, England
  - Southampton General Hospital, Southampton, England
  - South Warwickshire Hospital, Warwick, Warwickshire, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Royal Hampshire County Hospital, Winchester, England
  - Western Infirmary, Glasgow, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Hairmyres Hospital, Glasgow, Scotland
  - Crosshouse Hospital, Kilmarnock, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Withybush General Hospital, Haverfordwest, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales
  - South West Wales Cancer Institute, Swansea, Wales